CLINICAL TRIAL: NCT05967546
Title: Deep Learning for Intelligent Identification of Arrhythmias (ECG-LEARNING): an Investigator-initiated, National Multicenter, Retrospective-prospective, Cohort Study
Brief Title: Deep Learning for Intelligent Identification of Arrhythmias
Acronym: ECG-LEARNING
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: 521 Hospital of NORINCO Group (Other); Shaanxi Provincial People's Hospital (Other); Xiangyang Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2023LSK-170
Record Dates: First submitted 2023-07-06; First posted 2023-08-01 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Arrhythmia
Keywords: Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental Group: ECG data and clinical data from this group of arrhythmia patients will be used to build a deep learning model.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — No interventions will be given to patients.

SUMMARY:
This study aims to design and train a deep learning model for the diagnosis of different arrhythmias.

DETAILED DESCRIPTION:
This study aims to retrospectively and prospectively collect routine clinical data such as electrocardiograms from patients with arrhythmias who meet the inclusion and exclusion criteria. Then we will design and train a deep learning model to analyse the electrocardiographic features of the arrhythmias, and identify the types of arrhythmias and evaluate the value of the model for the diagnosis of different arrhythmias.

ELIGIBILITY:
Inclusion Criteria:

* For retrospective study: 1.Patients with arrhythmia diagnosed by routine surface 12-lead electrocardiogram or Holter; 2.The type of arrhythmia is diagnosed by intracardiac electrophysiological examination.
* For prospective study: 1.Patients with arrhythmia diagnosed by routine surface 12-lead electrocardiogram or Holter; 2.Intracardiac electrophysiological examination is planned.

Exclusion Criteria:

* Lack of routine surface 12-lead electrocardiogram or holter data;
* Lack of intracardiac electrophysiological examination;
* Patients refused to sign informed consent and refused to participate in the study.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with arrhythmia by twelve-lead electrocardiogram or Holter.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
A deep learning model designed to intelligently identify the types of arrhythmia. | 1 day after the enrollment.
  The model is trained on the training set, the best model and hyperparameters are selected through the verification set, and finally the model results are tested on the test set.

SECONDARY OUTCOMES:
The sensitivity, specificity and accuracy of the deep learning model | 1 day after the enrollment.
  The sensitivity, specificity and accuracy of a deep learning model designed were evaluated by intracardiac electrophysiological examination results to identify patients with arrhythmia from various centers.

CONTACTS AND LOCATIONS:
Overall Officials: Guoliang Li, M.D., Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiantong University, Xi'an, Shaanxi, China